CLINICAL TRIAL: NCT03807674
Title: A Prospective Clinical Pilot Study of MMP-9 Expression and Short-term Outcome of Coronal Pulpotomy in Mature Permanent Teeth With Symptomatic Pulpitis
Brief Title: MMP-9 Expression in Permanent Mature Teeth With Symptomatic Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eglė Gvazdaitytė (Other)
Responsible Party: Sponsor-Investigator, Eglė Gvazdaitytė, The senior resident of Lithuanian University of Health Sciences, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEC-LSMU(R)-01
Record Dates: First submitted 2018-11-19; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pulpitis
Keywords: Calcium-silicate, coronal pulpotomy, MMP-9, symptomatic pulpitis.
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group - Healthy teeth (Other): Patients with clinically healthy third molar or premolar teeth with indications for extraction; no clinical signs of pulpitis, no caries, no indications for the replacement of an old filling that is 1 mm from the pulp space as determined on the radiograph; a normal response to the cold test, and no apical radiolucency on the radiograph. For teeth of this group coronal pulpotomy was applied.
  Interventions: Procedure: Coronal pulpotomy
- Test group - Teeth with pulpitis (Experimental): Patients with symptomatic pulpitis resulting from caries; tooth pain defined as sharp, dull, localized or diffuse; pain at night; a symptomatic tooth with a positive response to the cold test and lingering pain; intermittent or continuous episodes of spontaneous pain (with no external stimulus) that could last from a few minutes up to a few hours; no apical radiolucency on the radiograph. For teeth of this group coronal pulpotomy was applied.
  Interventions: Procedure: Coronal pulpotomy

INTERVENTIONS:
Procedure: Coronal pulpotomy — Coronal pulpotomy was performed with a sterile high-speed round bur under water coolant. Pulp vitality was confirmed by the presence of bleeding pulp tissue from all of the canal orifices. Hemostasis was achieved through the application of a pellet moistened with 2.5% NaOCl for two minutes and was repeated as needed. Calcium-silicate based material was prepared ac-cording to the manufacturer's instructions and gently placed over the pulp to fill the entire cavity.

SUMMARY:
Matrix metallopeptidase-9 (MMP-9) expression was compared in healthy and inflamed pulp and the outcome of coronal pulpotomy in teeth with symptomatic pulpitis was assessed. After procedure blood samples were examined using Elisa kit.

DETAILED DESCRIPTION:
Introduction: Widely used diagnostic tests do not provide information to distinguish the pulp inflammation stage while improvement of materials, techniques and vital pulp therapy have received a wider acceptance in symptomatic pulpitis treatment. The aim of this clinical study was to compare MMP-9 expression in healthy and inflamed pulp and to assess the short-term outcome of coronal pulpotomy in mature permanent teeth with symptomatic pulpitis.

Methods: Patients diagnosed with symptomatic pulpitis were included in this clinical study. Coronal pulpotomy was performed using calcium-silicate based material and blood samples were taken. Initial and postoperative pain was recorded by Heft-Parker visual analog scale at 24 hours and 72 hours after the procedure. In control group teeth with healthy pulp were used. During follow-up visits after three and six-months, patients were examined clinically and radiographically. The ELISA kit was used to determine the levels of MMP-9 in inflamed and healthy coronal pulp tissue.

ELIGIBILITY:
Inclusion Criteria:

* Teeth diagnosed with symptomatic pulpitis
* Patients who did not use any NSAIDs before the treatment
* Positive cold test of investigated teeth
* Clinically dental caries in contact with pulp chamber
* Permanent teeth with radiographically closed root apex

Exclusion Criteria:

* Patients who refuse to participate in the study
* Medically compromised patients (with immunosuppressive/systemic diseases, patients on medications)
* Teeth with periapical radiolucency or clinical signs of apical periodontitis
* Periodontological compromised teeth (probing depth ≥4mm)
* Internal/external root resorption in periapical radiograph
* Pulp chamber and/or root canal calcification in periapical radiograph
* Teeth with unrestorable crown
* Teeth with a negative response to cold test

Ages: 14 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-02-11 (Actual)

PRIMARY OUTCOMES:
MMP-9 amount measurement using ELISA kit | All samples were measured in one time (during 12 hours)
  The MMP-9 amount in the pulp blood samples was measured using the MMP-9 Human ELISA Kit. The measurement procedure was followed according to the manufacturer's instructions. The anti-MMP-9 polyclonal antibody was pre-coated on 96-well plates. Blood samples and a biotin-conjugated antibody were added to the wells supplemented with Avidin-Biotin-Peroxidase Complex and 3,3',5,5'-tetramethylbenzidine in a mildly acidic buffer. A blue-colored product was produced and turned to yellow after an acidic stop solution was added. The intensity of the color yellow was proportional to the MMP-9 amount bound on the plate. The optical density absorbance was measured spectrophotometrically at 450nm in a microplate reader and the concentration of MMP-9 was calculated. For the expression of MMP-9 concentrations in the samples, a standard curve was used.

CONTACTS AND LOCATIONS:
Overall Officials: Greta Lodiene, Study Director — Lithuanian University of Health Science
Locations (1):
- Lithuanian University of Health Science, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided